CLINICAL TRIAL: NCT06512831
Title: Isoniazid Prophylaxis Based on Risk Factors of Tuberculosis in Living Kidney Transplantation Recipients: A Retrospective Cohort Study
Brief Title: Isoniazid Prophylaxis Based on Risk Factors of Tuberculosis in Living Kidney Transplantation Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Professor Tao Lin, West China Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WestChina-INH-KT
Record Dates: First submitted 2024-07-14; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplantation; Tuberculosis; Isoniazid Toxicity
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TB Risk factors with INH group (R-INH) (Experimental)
  Interventions: Drug: Isoniazid
- TB Risk factors without INH group (R-NINH) (No Intervention)
- Non-Risk group (NR) (No Intervention)

INTERVENTIONS:
Drug: Isoniazid — Those with risk factors were recommended a 6-month prophylaxis regimen, consisting of INH (300 mg/d) and pyridoxine (10 mg/d to prevent INH-related neurotoxicity).
  Arms: TB Risk factors with INH group (R-INH)

SUMMARY:
Tuberculosis (TB) is a major and severe opportunistic infection among solid organ transplant recipients. Chemoprophylaxis is advised for those with latent tuberculosis infection (LTBI). However, the effectiveness of an isoniazid (INH) prophylactic approach based on TB risk factors, without relying on tuberculin skin test (TST) or interferon-gamma release assay (IGRA), remains uncertain. Therefore, the investigators conducted this retrospective study to evaluate the safety and efficacy of a 6-month INH prophylaxis regimen guided by TB risk factors in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. living-donor kidney transplant recipients
2. receiving standard triad immunosuppressive regimen

Exclusion Criteria:

1. active TB infection
2. multiorgan transplantation
3. liver cirrhosis
4. malignancy history in the donor and recipient
5. human immunodeficiency virus infection
6. those who had received a nine-month course of INH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1348 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The incidence of post-transplant active TB | from transplant to post-transplant for up to 5 years

SECONDARY OUTCOMES:
The incidence of side effects of INH | Within 6 months of INH regimen

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No